CLINICAL TRIAL: NCT04077307
Title: A Phase 1 Study in Patients With Hematological Malignancies to Evaluate Safety, Tolerability and Efficacy of Karonudib
Brief Title: A Study in Leukemia Patients With Karonudib
Acronym: MAATEO
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Helleday Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MAATEO
Record Dates: First submitted 2019-08-26; First posted 2019-09-04 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Leukemia
Keywords: AML; ALL; MDS; Multiple myeloma; B cell lymphoma
MeSH Terms: conditions — Leukemia; Multiple Myeloma; Lymphoma, B-Cell | interventions — karonudib

STUDY DESIGN:
Intervention Model Description: First part of the study - 3 different dose cohorts with escalating doses are planned.
  Extension part of the study - 20 patients with diagnosis of Relapsed, Refractory or Progressive AML and MDS to be enrolled and treated with RP2D.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation (Experimental): Karonudib is an oral inhibitor of MTH1 and will be supplied as an oral solution to be taken every other day. There are three planned dose cohorts. Patients will be given every second day dosing.
  Interventions: Drug: Karonudib

INTERVENTIONS:
Drug: Karonudib — First part of the study - four different dose cohorts Extension part of the study - karonudib BID (twice a week) and Idarubicin days 1-3.

SUMMARY:
The primary objective of this study is to determine safety and tolerability of Karonudib for the treatment of hematological malignancies.

Secondary objectives are to determine a recommended RP2D and schedule for further development of Karonudib, to determine the pharmacokinetics of Karonudib, to look for evidence of treatment efficacy. Overall survival will also be recorded.

DETAILED DESCRIPTION:
Primary Objective Part I

* To determine the safety and tolerability of Karonudib in escalating doses for the treatment of patients with advanced relapsed/refractory Acute Myeloid Leukemia (AML), Acute Lymphoblastic Leukemia (ALL) , Diffuse Large B-Cell Lymphoma, Multiple Myeloma (MM) and high-risk Myelodysplastic Syndrome (MDS)AML, ALL, DLBCL, Burkitt´s lymphoma, multiple myeloma and high-risk MDS Primary Objective Part II
* To determine the safety and tolerability of Karonudib in combination with standard of care treatment, Idarubicinother anti-cancer agents for the treatment of patients with advanced progressive, relapsed/refractory AML, and high-risk MDS

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Age 18-75 years (may be extended to older if deemed fit).
3. The patient has received standard of care treatments and has refractory or relapsed or progressive disease with no suitable standard of care options available.

   For expansion cohort (Cohort V): Patients can only have received a maximum of 70% of anthracycline lifetime exposure to date of proposed dosing day.

   Cohorts I-IV: AML, ALL, DLBCL, Burkitt lymphoma, multiple myeloma or high-risk MDS, according to the WHO 2016 criteria.
4. Expansion cohort (Cohort V): Relapsed, Recurrent or Progressive AML or MDS according to the ELN 2017 criteriaWHO 2016 criteria.
5. For expansion cohort (Cohort V): Patients can only have received a maximum of 70% of anthracycline lifetime exposure to date of proposed dosing day.
6. The patient has received standard of care treatments and has refractory or relapsed disease with only experimental therapies as further treatment options.
7. Life expectancy of at least 8 weeks (as per investigators clinical assessment).
8. ECOG PFS 0-2
9. Patients must have measurable disease by blood or bone marrow or imaging examination.
10. Have a normal left ventricular ejection fraction (LVEF) based on institutional ranges.
11. Adequate hepatic and renal function defined as:

    1. Total bilirubin < 3 x ULN (does not apply to patients with Gilberts Syndrome).
    2. AST and ALT ≤ 5 x ULN.
    3. The calculated GFR is at least 30 ml/min using Cockcroft-Gault method.
12. Platelet count≥10 x 109/L. (Can be supported by platelet transfusion)
13. Subject must be able to take oral medication.
14. Negative pregnancy test according to CTFG guidance 2014 for females of child-producing potential.

Exclusion Criteria:

1. Age less than 18 years.
2. Less than 4 weeks since stopping previous systemic chemotherapy treatment with the exception of stable dose Hydroxyurea, Trophosphamide, oral Cyclophosphamide, ImID or Thioguanine which needs to be stopped 10 x t1/2 prior to Karonudib administration.
3. Less than 1 week since stopping palliative radiotherapy.
4. Less than 2 weeks after surgery except access surgical procedures.
5. Less than 6 months since a clinically significant cardiovascular event such as myocardial infarction, unstable angina, angioplasty, bypass surgery, stroke or TIA.
6. Congestive heart failure NYHA class > II.
7. History of arrhythmias or arrhythmias discovered during the screening period (apart from atrial fibrillation without ventricular tachycardia and premature extra beats).
8. Patients requiring anti-arrhythmic drugs except for stable dose beta-blocking or calcium channel blocking agents.
9. QTc interval >470 ms at baseline (Fridericia correction).
10. Use of Fentanyl (must be stopped at least 1 week prior to initiation of Karonudib).
11. Use of anti-oxidants vitamins and Acetylcysteine (must be stopped within 48 hours of starting treatment with Karonudib).
12. Use of antidepressant medications which are substrate for CYP2D6 (must be stopped at least 3 weeks prior to starting treatment with Karonudib).
13. Any severe acute or chronic medical condition that places the patient at increased risk or interferes with the interpretation of study results.
14. Intracerebral engagement (patient with previously known engagement are eligible provided that there is no evidence of disease progression for a minimum of 8 weeks prior to inclusion.
15. Known acute or chronic infection with hepatitis B or C except for DNA-negative hepatitis B with stable dose anti-viral agents.
16. Known HIV infection.
17. Pregnant or breast-feeding women.
18. Patients with reproductive potential not implementing accepted and effective means of contraception.
19. Participation in any other clinical trial with a pharmaceutical product within 5 x t½, or minimum 1 week, since last dosing of the IMP, whichever is the shorter.
20. Acute promyelocytic leukemia (AML M3).
21. Uncontrolled ongoing systemic or localized infection.
22. Unable to comply with study procedures.
23. Peripheral neurological toxicity CTCAE grade 2 or higher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2019-12-03 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety of Karonudib (TH1579) | 28 days, first treatment cycle for the patient.
  Grade and frequency of AE and SAE using the CTCAE version 5.0
Tolerability of Karonudib (TH1579) | 28 days, first treatment cycle for the patient.
  Grade and frequency of AE and SAE using the CTCAE version 5.0

SECONDARY OUTCOMES:
Preliminary signs of clinical efficacy of Karonudib. | 28 days, first treatment cycle for the patient.
  ELN/IWG response criteria

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Deneberg, MD, Principal Investigator — Karolinska University Hospital
Locations (6):
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet Copenhagen University Hospital, Copenhagen
- Serbia (2):
  - University Clinical Center Belgrade, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
- Sweden (2):
  - Karolinska University Hospital, Huddinge
  - Örebro University Hospital, Örebro

IPD SHARING:
Plan to Share IPD: No